CLINICAL TRIAL: NCT01505660
Title: Randomized Controlled Trial Using Patient Reported Outcomes and Care Managers to Improve HIV Medication Adherence in Routine Clinical Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Heidi Crane, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Purpose: Supportive Care
Other Study IDs: 41128-K; R01MH084759 (NIH); U01AR057954 (NIH); ADH HIV001 (Other: UW)
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: HIV
Keywords: Adherence; Depression; Care management; Stepped care; HIV; Patient reported outcomes; Antiretroviral medication adherence
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Patients not randomized to the intervention will receive usual care which includes a patient reported outcomes assessment every 6 months as part of routine clinical procedures and patient-initiated interactions with case managers.
- Care management (Experimental): The intervention will include frequent healthcare delivery team notification of PROs including medication adherence and adherence barriers such as depression symptoms along with tailored intervention recommendations and targeted care management using a stepped care approach.
  Interventions: Behavioral: Care management

INTERVENTIONS:
Behavioral: Care management — The intervention will include healthcare delivery team notification of patient reported outcomes (PROs) including medication adherence and adherence barriers such as depression symptoms along with intervention recommendations and targeted care management using a stepped care approach. Patients will receive structured calls from their care manager 2 and 6 weeks after enrollment. An assessment including depression, adherence, and substance use will be completed at the beginning of each call. After the 2nd call, a stepped care approach will be used where patients with a greater need based on adherence and depression will receive more intensive interventions based on the PEARL intervention. The components include: a) problem solving treatment, b) social and physical activation, c) pleasant events scheduling, d) patient support and education regarding medication use, and e) medical and psychiatric consultation. Patients will also receive follow-up calls at ~9 and 12 months after enrollment.
  Arms: Care management

SUMMARY:
Among HIV-infected patients, adherence to antiretroviral medications is one of the most important determinants of clinical outcomes including viral suppression, viral resistance, disease progression, and death. Unfortunately poor adherence among patients with HIV is very common, mean levels of adherence in clinical cohorts are 60-75% or less. Alcohol, drug abuse, and mental illness particularly depression symptoms are key predictors of poor adherence, common among HIV-infected individuals, and important to identify and treat among nonadherent patients. This study will examine the ability of patient reported outcomes (PROs) and a targeted care management approach to improve clinical outcomes with a randomized controlled trial (RCT) in routine clinical care of patients with HIV. The investigators will determine whether healthcare delivery team notification of PROs including antiretroviral medication adherence and barriers of adherence such as depression and substance abuse along with tailored intervention recommendations and targeted care management leads to improvement in both process and clinical outcomes including patient-reported outcomes. The investigators will examine process outcomes such as use of clinic support services, and patient outcomes such as improvement in adherence, substance use, depression, and HIV-1 RNA levels.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individuals
* English speaking
* 18 years of age or older
* Access to either a home phone or cell phone at enrollment
* In care at least 6 months.
* Self-reported inadequate adherence based on routine clinic assessment

Exclusion Criteria:

* Do not speak English
* Not receiving antiretroviral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Self-reported adherence | up to 1 year after enrollment

SECONDARY OUTCOMES:
HIV-1 RNA level | up to 1 year after enrollment
Self-reported substance use | Up to 1 year after enrollment
Health related quality of life | Up to 1 year after enrollment
Physical activity levels | up to 1 year after enrollment
Self-reported depression | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M Crane, MD, MPH, Principal Investigator — University of Washington; Paul K Crane, MD MPH, Principal Investigator — University of Washington; Donald Patrick, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Crane HM, Fredericksen RJ, Church A, Harrington A, Ciechanowski P, Magnani J, Nasby K, Brown T, Dhanireddy S, Harrington RD, Lober WB, Simoni J, Safren SA, Edwards TC, Patrick DL, Saag MS, Crane PK, Kitahata MM. A Randomized Controlled Trial Protocol to Evaluate the Effectiveness of an Integrated Care Management Approach to Improve Adherence Among HIV-Infected Patients in Routine Clinical Care: Rationale and Design. JMIR Res Protoc. 2016 Oct 5;5(4):e156. doi: 10.2196/resprot.5492. PMID 27707688